CLINICAL TRIAL: NCT01174914
Title: Phase 2 Comparison of Low-Dose Naltrexone vs ARV Effectiveness in HIV+ Progression
Brief Title: Effectiveness Study Low-Dose Naltrexone Versus ARV's for HIV+
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Ojai Foundation (Other)
Responsible Party: Abdel Kader Traore, MD, PI, Professor Bamako University School of Medicine, Pharmacy and Odontostomatology, University of Bamako (Mali) Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TOFLDNMALIHIVb
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: HIV Seropositivity
MeSH Terms: conditions — HIV Seropositivity | interventions — Lamivudine; Nevirapine; Stavudine; stavudine, lamivudine, nevirapine drug combination; efavirenz; Emtricitabine; Tenofovir; Naltrexone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Naltrexone Low-dose 3mg capsule (Experimental): Each person in this arm 1 of the study had never received any ARV drugs and in this study received only one Low-Dose Naltrexone 3mg capsule nightly for 9 months (no placebo).
  Interventions: Drug: Naltrexone
- Naltrexone Low Dose + ARVs (Active Comparator): In this Arm 3, Patients were on ARV's plus being given Naltrexone Low-Dose (3mg) once daily at bedtime for 9 months.
  Interventions: Drug: Naltrexone + ARV's
- ARV's (continued,standard) plus Placebo (Placebo Comparator): In this arm 2, patients were started or continued on their standard ARV drugs plus placebo capsule once daily at bedtime; in the 2nd and 3rd arms patients did not know whether they were taking Low-Dose Naltrexone or a placebo.
  Interventions: Other: ARV's + Placebo

INTERVENTIONS:
Other: ARV's + Placebo — Patients continued ARV's plus a placebo nightly for 9 months
  Other Names: Azidothimidine + lamivudine + nevirapine Or; Stavudine + lamivudine + nevirapine (TRIOMUNE)Or; Azidothimidine + lamivudine + efavirenz Or; Azidothimidine + lamivudine + lopinavir/r Or; Emtricitabine + tenofovir + efavirenz
  Arms: ARV's (continued,standard) plus Placebo
Drug: Naltrexone — Naltrexone, Low-Dose (3mg) given once daily at bedtime for 9 months
  Arms: Naltrexone Low-dose 3mg capsule
Drug: Naltrexone + ARV's — Patients were given standard ARV's plus Naltrexone (Low Dose) 3mg nightly.
  Other Names: Azidothimidine + lamivudine + nevirapine Or; Stavudine + lamivudine + nevirapine (TRIOMUNE)Or; Azidothimidine + lamivudine + efavirenz Or; Azidothimidine + lamivudine + lopinavir/r Or; Emtricitabine + tenofovir + efavirenz
  Arms: Naltrexone Low Dose + ARVs

SUMMARY:
In the vast majority of those infected with HIV virus who are untreated, there is deterioration in immune health over a period of months or years inevitably leading to full-blown AIDS and demise. Treatment with ARV's stop or slow down this deterioration if started before a certain degree of progression occurs and has saved millions of lives. The investigators' study hypothesis is that effectiveness of a very low dose of an FDA-approved medication, naltrexone hydrochloride, (Low-Dose Naltrexone, or LDN) will compare favorably to ARV's to prevent progression of HIV+ toward immune deterioration and full-blown AIDS.

DETAILED DESCRIPTION:
The LDN (low-dose naltrexone) vs ARV (anti-retroviral drugs) Effectiveness Study in Mali sponsored by The Ojai Foundation in California-USA is a clinical research study endorsed and approved by the Malian Government. Naltrexone hydrochloride is a generic, FDA-approved since 1998 drug, an opioid antagonist that has clinically shown immune enhancing/modulating qualities in very low dosage and may offer an alternative to ARV drugs that is effective, non-toxic, easily available, inexpensive, with simple once-daily at bedtime administration. LDN capsules must be created by compounding pharmacists to get these ultra-small doses. Due to toxicity of current ARV drugs and need for special medical management young HIV infected children are largely neglected particularly in developing countries; LDN can also be made available in a transdermal cream for infants and children who are HIV infected.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* CD4 count over 350 (arm 1/group 1)
* CD4 count over 200 and on ARV's (arms 2,3/groups 2,3)
* Age between 18 & 60
* Males or females

Exclusion criteria:

* HIV-1 seronegative
* HIV-2 infected
* CD4 count lower than 200
* patients under age 18
* Those refusing to be in study
* Pregnant or breast-feeding women
* Patients under immuno-suppressor therapy
* Those with renal or hepatic dysfunction
* Malaria or tuberculosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
CD4+ percentage (change in HIV-1 seropositive patients) | 9 MONTHS
  HIV+ patients with CD4+ count over 350 had their CD4 count/percentage measured at beginning, at 15 days, at 1 month, 3 months, 6 months and 9 months (end).

SECONDARY OUTCOMES:
Clinical assessment of evidence of AIDS or other serious illness | 9 MONTHS
  HIV+ patients with CD4 counts over 200 on ARV drugs were given clinical assessment and testing for evidence of opportunistic infections (AIDS) at each visit for blood testing: (Beginning, 15 days, 1 month, 3 months, 6 months, & 9 months (end).

CONTACTS AND LOCATIONS:
Overall Officials: Abdel K Traore, MD, Principal Investigator — Professor, Bamako University School of Medicine
Locations (1):
- University Hospital of Point G, Bamako, Mali